CLINICAL TRIAL: NCT05577351
Title: PULSE-F: Feasibility Study of RapidPulseTM Aspiration System as Frontline Approach for Patients With Acute Ischemic Stroke Due to Large Vessel Occlusions
Brief Title: Feasibility Study of RapidPulseTM Aspiration System as Frontline Approach for Patients With Acute Ischemic Stroke
Acronym: PULSE-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RapidPulse, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-0004
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Large Vessel Occlusion; Mechanical Thrombectomy; Neurovascular Intervention
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Thrombectomy

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, open-label, single-arm study to assess the initial technical effectiveness and safety of the RapidPulseTM (feasibility version). As such, no formal statistical hypothesis will be tested in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Each subject will undergo baseline evaluation for acute ischemic stroke due to large vessel occlusion, per standard of care and undergo mechanical thrombectomy procedure, aspiration to remove thrombus in the neuro-vasculature using the RapidPulseTM (feasibility) device.
  Interventions: Device: RapidPulseTM Aspiration System

INTERVENTIONS:
Device: RapidPulseTM Aspiration System — The RapidPulseTM Aspiration System paired with a single-use, disposable tubing set specific for use with the RapidPulseTM Aspiration System
  Other Names: Aspiration Thrombectomy

SUMMARY:
A feasibility study to evaluate the initial safety and performance of the RapidPulseTM Aspiration System in the treatment of patients with Acute Ischemic Stroke (AIS) due to Large Vessel Occlusion (LVO) in the intracranial ICA, M1, M2, basilar or vertebral arteries.

DETAILED DESCRIPTION:
The purpose of this prospective, open label clinical trial is to assess the initial safety and performance of the RapidPulseTM Aspiration System as frontline approach for patients with acute ischemic stroke due to large vessel occlusions identified within 24 hours of symptom onset (or last seen normal). The study will enroll up to a maximum of 50 subjects in 2 centers in Georgia. Subjects will undergo mechanical thrombectomy procedure and will have post-operative assessments completed at 24 hours and on Day 5-7 or upon hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of acute ischemic stroke with symptom onset (or last seen normal) within 24 hours
* Large vessel occlusion (LVO) involving the intracranial internal carotid artery (ICA), middle cerebral artery (MCA) M1 or M2 segments, basilar or vertebral artery
* Target occlusion can be accessed by the Medtronic React 71 aspiration catheter

Exclusion Criteria:

* Known or suspected intracranial atherosclerotic disease (ICAD)
* Tandem occlusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
First Pass Reperfusion Effect (FPE) | Intra-procedural
  Defined by mTICI greater than or equal to 2c after one reperfusion attempt

OTHER OUTCOMES:
Frontline Technical Success | Intra-procedural
  As defined by mTICI 2b or greater after the last pass with Study Device (no rescue therapy)
Final mTICI | Intra-procedural
  After all passes (including any rescue therapy)
Modified First Pass Reperfusion Effect (mFPE) | Intra-procedural
  Defined as mTICI 2b or greater after one device pass
Device-related and procedure-related adverse events | Intra and post-procedural (up to 24 hours)
  Including vessel injury, distal emboli, emboli in new territory (ENT) and vessel spasm

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Study Chair — University of Pittsburgh Medical Center Stroke Institute
Locations (2):
- Georgia (2):
  - National Institute of Surgery, Tbilisi
  - Pineo Medical Ecosystems, Tbilisi

IPD SHARING:
Plan to Share IPD: No